CLINICAL TRIAL: NCT05248854
Title: Effects of Sensorimotor and Core Stabilization Exercise Programs Following Total Knee Arthroplasty : A Randomize Controlled Trial
Brief Title: Effects of Sensorimotor and Core Stabilization Exercises After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YeditepeUPT
Record Dates: First submitted 2022-01-11; First posted 2022-02-21 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis; Arthroplasty; Joint Replacement
Keywords: total knee replacement; arthroplasty; balance; core stabilization; sensorimotor training
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial , prospective, single bllinded.
Who Masked: Participant
Masking Description: Participants did not know the their grup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor exercise training (Experimental): SM program included combination of traditional hip and knee exercise, various balance and proprioceptive exercises.
  Interventions: Other: Sensorimotor exercise training
- Core Stabilization exercise training (Experimental): Core stabilization exercise program contained traditional hip and knee ROM exercise combining the core stabilization as mat activities
  Interventions: Other: Core stabilization exercise training

INTERVENTIONS:
Other: Sensorimotor exercise training — The program included side stepping, tandem walking, perturbation exercise, overcoming mini obstacles, walking different surfaces and traditional hip and knee exercise. Participants applied these exercise as home program between postoperative second weeks and 8th weeks, 3-5 day /week , 20 25 min every session.
  Other Names: SM exercises
  Arms: Sensorimotor exercise training
Other: Core stabilization exercise training — Core stabilization exercise program was also prepared parallel to the sensorimotor training group intensity; the program contained traditional hip and knee exercise combining the core stabilization as mat activities depending on previous research.core stabilization exercise program was also prepared parallel to the sensorimotor training group intensity; the program contained traditional hip and knee exercise combining the core stabilization as mat activities depending on previous research
  Other Names: CS exercises
  Arms: Core Stabilization exercise training

SUMMARY:
Tha aim of the study is to investigate the effects of core stabilization and sensorimotor exercise program on range of motion, proprioception, balance and functional status in patients with total knee arthroplasty. The study lasts prospective randomized controlled trial. Participants were randomly divided into sensorimotor training (SM,n=17) and core stabilization training group (CS,n=19). The exercise training program was administered for home exercise as 3-5 times a week and for a 6-week duration.

DETAILED DESCRIPTION:
Objective :

To investigate the effects of core stabilization and sensorimotor exercise program on range of motion, proprioception, balance and functional status in patients with total knee arthroplasty.

Design :

Prospective randomized controlled trial

Subjects :

A total of 36 Ostearthritis patients (69.8 ± 5.1 years) who underwent unilateral knee arthroplasty. Participants were performed TKA surgery by the same physician and followed by the same therapist.

The following inclusion criteria were used: being volunteer, 50-85 age range, being diagnosed with stage 4 OA and undergoing unilateral TKA surgery. The following exclusion criteria were applied: having previous surgery history of affected lower limb, impaired hearing, vision or verbal problems, physical or mental disability, having a neurological or oncologic disease that may affect functional performance.

Patients who met inclusion criteria and were willing to join the study (n=52) were evaluated after being diagnosed with OA and before the operation at the clinic. A total 40 patients undergoing TKA surgery participated in our study and were randomly separated to the Sensorimotor Training Group (SM, n=20) and the Core Stabilization Training Group (CS, n=20). Group allocation was randomized in two blocks of 40 sealed envelopes without external marks, which were mixed and numbered from 1 to 40, containing a piece of paper with the group allocation. All participants were blinded to the treatment type. As a result, 36 patients completed the process.

Outcome Measures :

Patients were assessed on three separate occasions (presurgery, 2 weeks and 8 weeks postsurgery). The primary outcome was proprioception and seconder outcomes were range of motion, Knee Injury and Osteoarthritis Outcome Scale (KOOS), Berg Balance Test, Timed-up & Go test and Sit & Stand -Up tests.

Interventions :

Participants were randomized into two intervention groups: sensorimotor training group (SM, n=17) and Core Stabilization training group (CS, n=19). Both groups were prescribed a 6-week home based exercise programme for 3-5 sessions/week between 2 and 8 weeks postsurgery.

ELIGIBILITY:
Inclusion Criteria:

* being volunteer,
* 50-85 age range,
* being diagnosed with unilateral OA and undergoing unilateral TKA surgery

Exclusion Criteria:

* having previous surgery history of lower limbs,
* impaired hearing-vision -verbal problems, physical or mental disability,
* having a neurological or oncologic disease that may affect functional performance.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Proprioception | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  Joint Position Sense(JPS) was assessed to proprioception. JPS was evaluated via ability to reproduce joint angles using position-matching with active or passive movements (21, 22). Therapist showed each reference 30 and 60 degree flexion angles passively three times, held it for 10 second and returned to starting position during sitting. Then, patients were asked to show the target angles with eyes-closed, three deviated angles were recorded and the mean of errors was used for statistics

SECONDARY OUTCOMES:
Range of motion (ROM) | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  The ROM of knee and hip joints were assessed bilaterally via a universal goniometer.
Sit to Stand Test | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  The STS test was applied by recording the elapsed time between the patients who were asked to sit and stand up 5 times as fast as possible
Timed up and Go Test | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  In the TUG test, patients were asked to stand up independently from the chair, walk 3 m, turn around and sit at the starting point; the time elapsed between them was recorded (25). The minimum 2.49 seconds change indicates good clinical properties and below the 14 sec during performance indicate higher risk of falling.
Berg Balance Test | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  Berg Balance Test was also used to assess the static balance and falling risk of the participants. The test includes 14 different tasks scored between 0-4 points. Total scores were recorded between 0-56 points, higher score indicates better balance level
KOOS Scale | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  KOOS consists of 42 items and five subscales: pain, symptom, activities of daily life, quality of life, sport and recreation. All questions are scored 0-4 points and subscales points are converted separately to 0-100 points. Higher point indicates no knee problems
Tampa Scale of Kinesiophobia | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  Consist of 17 items, evaluate the fear of movement.
Oswestry Low Back Disability Questionnaire | change from baseline to postsurgery second weeks , change from postsurgery second weeks to eighth weeks
  The Oswestry Disability Index is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah DEMİRBAŞ, Operator, Study Chair — Tuzla Gispir Hospital; Şule BADILLI HANTAL, PhD, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)